CLINICAL TRIAL: NCT01841632
Title: Safety and Feasibility of Multipotent Adult Progenitor Cells for Immunomodulation Therapy After Liver Transplantation: A Phase I Study of the MiSOT Study Consortium
Brief Title: Safety Study of Multipotent Progenitor Cells for Immunomodulation Therapy After Liver Transplantation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Prof. Dr. Marc-H. Dahlke, Ph. D. (Other)
Collaborators: University Hospital Regensburg (Other); Healios K.K. (Industry)
Responsible Party: Sponsor-Investigator, Prof. Dr. Marc-H. Dahlke, Ph. D., Sponsor-Investigator, University Hospital Regensburg
Organization: University Hospital Regensburg (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MISOT-I; 2009-017795-25 (EudraCT Number)
Record Dates: First submitted 2013-04-19; First posted 2013-04-26 (Estimated); Results first posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2017-12

CONDITIONS: Liver Transplantation
Keywords: Liver transplantation; Allogeneic liver transplantation; Solid organ transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MultiStem (Experimental): Dose escalation
  Cohort 1
  Drug: MultiStem, Dose 1 of MultiStem; Route and time: Two infusions; First: intra portal at liver transplantation (day 1), second: intra venous (day 3)
  Cohort 2
  Drug: MultiStem, Dose 2 of MultiStem; Route and time: Two infusions; First: intra portal at liver transplantation (day 1), second: intra venous (day 3)
  Cohort 3
  Drug: MultiStem, Dose 3 of MultiStem; Route and time: Two infusions; First: intra portal at liver transplantation (day 1), second: intra venous (day 3)
  Cohort 4
  Drug: MultiStem, Dose 4 of MultiStem; Route and time: Two infusions; First: intra portal at liver transplantation (day 1), second: intra venous (day 3)
  Interventions: Drug: MultiStem

INTERVENTIONS:
Drug: MultiStem

SUMMARY:
MultiStem ® is a new biological product, manufactured from human stem cells obtained from adult bone marrow. Factors expressed by MultiStem cells are believed to regulate immune system function and augment tissue repair.

Standard of care pharmacological immunosuppression after liver transplantation can achieve reasonable survival of liver grafts and patients. The side effects of this treatment, however, are clinically significant and diminish the overall success of organ transplantation as a curative therapy. It is therefore the objective of this study to implement cellular immunomodulation therapy with MultiStem as an adjunct to standard pharmacological immunosuppression with the ultimate goal of significantly reducing drug-based immunosuppression.

As this is the first study with MultiStem in this subject population it has been designed as a safety and feasibility trial. However, first evidence of a potential benefit for this patient population will be explored cautiously.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age undergoing allogeneic liver transplantation
* Absence of any familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Written informed consent prior to any study procedures

Exclusion Criteria:

* Known allergies to bovine or porcine products or any other ingredients of the product
* Patients older than 65 years of age
* Patients listed in a high-urgency status that would not allow proper preparation of the study interventions
* Patients receiving a secondary liver graft (Re-Transplantation)
* Double organ transplant recipients
* Pre-existing renal failure that requires or has required hemodialysis within the last year
* Pulmonary function: FEV1, FVC, DLCO ≤50% predicted
* Cardiac function: left ventricular ejection fraction ≤50%
* HIV seropositive, varicella virus active infection or any other clinically relevant infection
* History of any malignancy (including lymphoproliferative disease and hepatocellular carcinoma) except for squamous or basal cell carcinoma of the skin that has been treated with no evidence of recurrence
* Unstable myocardium (evolving myocardial infarction), cardiogenic shock
* Females of childbearing potential (hormonal status and gynecological consultation required)
* Patients with portal vein thrombosis
* Patients with a history of pulmonary embolism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, University Hospital Regensburg, Regensburg, Bavaria, Germany

REFERENCES:
- [Background] Popp FC, Fillenberg B, Eggenhofer E, Renner P, Dillmann J, Benseler V, Schnitzbauer AA, Hutchinson J, Deans R, Ladenheim D, Graveen CA, Zeman F, Koller M, Hoogduijn MJ, Geissler EK, Schlitt HJ, Dahlke MH. Safety and feasibility of third-party multipotent adult progenitor cells for immunomodulation therapy after liver transplantation--a phase I study (MISOT-I). J Transl Med. 2011 Jul 28;9:124. doi: 10.1186/1479-5876-9-124. PMID 21798013
- [Background] Dillmann J, Popp FC, Fillenberg B, Zeman F, Eggenhofer E, Farkas S, Scherer MN, Koller M, Geissler EK, Deans R, Ladenheim D, Loss M, Schlitt HJ, Dahlke MH. Treatment-emergent adverse events after infusion of adherent stem cells: the MiSOT-I score for solid organ transplantation. Trials. 2012 Nov 15;13:211. doi: 10.1186/1745-6215-13-211. PMID 23151227

RESULTS

PARTICIPANT FLOW:
Groups:
- MultiStem - Cohort 1: Cohort 1
  Drug: MultiStem, Dose 1 of MultiStem; Route and time: Two infusions; First: intra portal at liver transplantation (day 1), second: intra venous (day 3)
Period: Overall Study
Arm/Group | MultiStem - Cohort 1
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MultiStem - Cohort 1
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  Germany | 3

OUTCOME MEASURES:

1. Primary Outcome: Infusional and Acute Toxicity, Using Toxicity Scoring Mechanism
Description: * For the description of intraportal toxicity a doppler ultrasound examination will be performed to assess various parameters that describe velocity of flow and flow pattern.
  * For pulmonary toxicity the assessment begins with an arterial blood gas. If this reveals pathological findings, a chest X-ray is required for clinical reasons independent of the study enrolment. In addition, clinical data describing the need for postoperative re-intubation will be recorded and the patient is assessed for the occurrence of a pulmonary embolism according to clinical guidelines.
  * For systemic toxicity, the occurrence of anaphylactic shock due to standard clinical guidelines is recorded.
Time Frame: up to day 30 (+10)
Population: A Per-protocol (PP) population consisting of all patients of the ITT population who showed no major protocol violations.
Measure: Count of Participants; unit: Participants
Arm/Group | MultiStem - Cohort 1
Number analyzed (Participants) | 3
Participants | 0

2. Secondary Outcome: Time to First Biopsy-proven Acute Rejection
Description: Per protocol biopsies will be performed on days 1, 4, 10. Additional biopsies will be taken whenever clinically necessary.
Time Frame: up to day 90 (+/-30)
Reporting Status: Not Posted

3. Secondary Outcome: Evidence Confirming That MultiStem Does Not Promote Malignant Transformation or Tumor Growth
Description: Four additional outpatient visits are planned to further evaluate the study patients (including screening for malignancies).
Time Frame: up to day 365 (+/-30)
Population: A Per-protocol (PP) population consisting of all patients of the ITT population who showed no major protocol violations. Protocol violations that may have an impact on the study outcome were considered as major protocol violations.
Measure: Count of Participants; unit: Participants
Arm/Group | MultiStem - Cohort 1
Number analyzed (Participants) | 3
Participants | 0

4. Secondary Outcome: Evaluation of Data From Routine Examinations Following Last Study Visit for Evidence of Long Term Safety From MultiStem Administration
Description: The results of routine examinations, which are necessary for all transplant patients, will be used once a year and analyzed retrospectively.
Time Frame: up to six years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The period of (S)AE reported for each trial patient was from the time of first study-specific procedure until 30 days after the final trial visit (approximately 52 weeks) or until the date of patient withdrawal.
Arm/Group | MultiStem - Cohort 1
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MultiStem - Cohort 1 (N=3)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 2 (3)
Liver function test abnormal (Investigations) | 1 (1) — abnormal AST, ALT and bilirubin values
Liver transplant rejection (Immune system disorders) | 1 (1) — acute rejection
Papilla of Vater stenosis (Gastrointestinal disorders) | 1 (1) — stenosis of papilla duodeni major
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MultiStem - Cohort 1 (N=3)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Abnormal faeces (Gastrointestinal disorders) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Agitation (Psychiatric disorders) | 2 (5)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dysphemia (Psychiatric disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Impaired healing (General disorders) | 2 (2)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Infection (Infections and infestations) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (2)
Liver function test abnormal (Investigations) | 2 (2)
Myopia (Eye disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (4)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Oedema (General disorders) | 1 (2)
Oedema peripheral (General disorders) | 1 (2)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Oropharyngeal pain (Gastrointestinal disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal function test abnormal (Investigations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Wound infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes